CLINICAL TRIAL: NCT04406727
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Trial With UB-421 in Combination With Optimized Background Regimen in Patients With Multi-drug Resistant HIV-1 Infection
Brief Title: UB-421 in Combination With Optimized Background Regimen in Patients With Multi-drug Resistant HIV-1 Infection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBP-A308-HIV
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — UB-421; Anti-Retroviral Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UB-421 (Experimental): 2-arm Comparison Phase: UB-421(25 mg/kg, every 2 weeks) in combination with ARV
  Single-arm Maintenance Phase: UB-421 plus optimized background regimen (OBR).
  Interventions: Biological: UB-421; Other: Antiretroviral (ARV)
- Placebo (Active Comparator): 2-arm Comparison Phase: Placebo in combination with ARV
  Single-arm Maintenance Phase: UB-421 plus optimized background regimen (OBR).
  Interventions: Other: Antiretroviral (ARV)

INTERVENTIONS:
Biological: UB-421 — UB-421 in combination with their ARV
  Arms: UB-421
Other: Antiretroviral (ARV) — Antiretroviral (ARV)

SUMMARY:
The purpose of this phase III study is to evaluate the efficacy between treatments (UB-421 Arm vs. Placebo Arm) by measuring the proportion of subjects with reduction in HIV-1 RNA viral load.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 seropositive
2. Have a history of at least 6 months on antiretroviral treatment
3. Receiving a stable combination antiretroviral therapy (ART) for at least 8 weeks before Screening

Exclusion Criteria:

1. Subjects with HBsAg positive or HCV antibody positive, along with ALT or AST > 4 x upper limit of normal (ULN)
2. Females who are pregnant
3. Any vaccination within 2 weeks prior to the Screening
4. Any prior exposure to UB-421

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HIV-1 RNA viral load between 2 arms | 14 Days